CLINICAL TRIAL: NCT02363439
Title: An Extension Study to Evaluate the Long-Term Safety, Tolerability, and Clinical Activity of IMO-8400 in Patients With Relapsed or Refractory Waldenström's Macroglobulinemia Who Completed Study 8400-401
Brief Title: Extension Study of IMO-8400 in Patients With Waldenström's Macroglobulinemia Who Completed Study 8400-401
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8400-404
Record Dates: First submitted 2014-11-19; First posted 2015-02-16 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — bazlitoran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg 2xwk (Experimental): Subcutaneous injection of IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg twice weekly per Protocol 8400-401
  Interventions: Drug: IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg twice weekly

INTERVENTIONS:
Drug: IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg twice weekly — IMO-8400 at 0.6 mg/kg/wk or 1.2 mg/kg twice weekly as defined per Protocol 8400-401

SUMMARY:
An extension study for patients who complete 24 weeks of IMO-8400 on study 8400-401.

DETAILED DESCRIPTION:
Patients who had no evidence of disease progression or toxicity while participating in study 8400-401 (NCT02092909) will continue to receive IMO-8400 until disease progression, adverse event or the investigator deems the goals of extended treatment with IMO-8400 have been met.

ELIGIBILITY:
Inclusion Criteria:

* Completed 24 weeks of treatment in Protocol 8400-401

Exclusion Criteria:

* Grade 3 (or higher) adverse event assessed as treatment-related at any time during the course of treatment under Protocol 8400-401.
* Has evidence of disease progression under Protocol 8400-401.
* Has received other anti-cancer therapies other than IMO-8400 since enrolling in Protocol 8400-401.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cornfeld, MD, MPH, Study Director — Idera Pharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg 2xwk
Started | 5
Completed | 1
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg 2xwk: Subcutaneous injection of IMO-8400 0.6 mg/kg/wk or 1.2 twice weekly per Protocol 8400-401
Arm/Group | IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg 2xwk
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Long term safety and tolerability of IMO-8400 in patients with Waldenstrom's Macroglobulinemia
Time Frame: During receipt of study treatment on the trial.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | IMO-8400 0.6 mg/kg/wk or 1.2 mg/kg 2xwk
Number analyzed (Participants) | 5
Participants | 4

ADVERSE EVENTS:
Time Frame: During receipt of study treatment on the trial.
Description: An Adverse Event is any untoward medical occurrence temporally associated with the use of a medical product in a patient, whether or not the event is considered causally related to the medical product.26 An AE can be a new occurrence or an existing process that increases significantly in intensity or frequency.
Groups:
- IMO-8400 at 0.6 mg/kg/wk or 1.2 mg/kg 2xwk: Subcutaneous injection of IMO-8400 0.6mg/kg/wk or 1.2 mg/kg twice weekly per Protocol 8400-401
Arm/Group | IMO-8400 at 0.6 mg/kg/wk or 1.2 mg/kg 2xwk
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMO-8400 at 0.6 mg/kg/wk or 1.2 mg/kg 2xwk (N=5)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Conjunctival hemorrhage (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site bruising (General disorders) | 1
Injection site discoloration (General disorders) | 1
Injection site erythema (General disorders) | 1
Edema peripheral (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes